CLINICAL TRIAL: NCT03240081
Title: Treating Where it Hurts: A Randomized Blinded Clinical Trial of Local Estrogen to the Vulvar Vestibule for Dyspareunia in Postmenopausal Women
Brief Title: Treating Postmenopausal Dyspareunia Where it Hurts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OHSU IRB 16770
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Dyspareunia
Keywords: Post-menopause dyspareunia; Vulvar vestibular pain; Genitourinary syndrome of menopause; Sexual pain
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50mcg estradiol cream (Active Comparator): Subjects randomized to 50mcg of study medication will be issued a pump that will dispense 0.5gm of cream with each pump
  Interventions: Drug: 50mcg estradiol cream
- 100mcg estradiol cream (Active Comparator): Subjects randomized to 100mcg of study medication will be issued a pump that will dispense 0.5gm of cream with each pump
  Interventions: Drug: 100mcg estradiol cream

INTERVENTIONS:
Drug: 50mcg estradiol cream — Use of study drug nightly applied to vulvar vestibule
  Arms: 50mcg estradiol cream
Drug: 100mcg estradiol cream — Use of study drug nightly
  Arms: 100mcg estradiol cream

SUMMARY:
The purpose of this study is to compare the effectiveness of two low doses of estrogen cream applied to a new location for the treatment of moderate or severe pain during sexual intercourse in postmenopausal women.

DETAILED DESCRIPTION:
Estrogen cream is FDA-approved for vaginal use for the treatment of sexual pain, but its use in a new location is experimental. Pain with sex is a common problem experienced by women after menopause and the relationship of pain to sexual difficulties is well established. The cause has been assumed to be atrophy and the location has been assumed to be the vagina. Recent focused studies have shown that the location of pain is the vulvar vestibule and usually not the vagina. This study will look at pain before and after therapy with estrogen when only the vulvar entryway area is treated. This will be a study focused on sexual dysfunction in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women aged 40 to 70 years old.
2. Postmenopausal, demonstrated by at least one of the following:

   i. Cessation of menses for ≥1 years if age is >50 ii. Bilateral oophorectomy iii. A history of climacteric symptoms if below age 50, having an ovary and scarred or absent uterus.
3. Onset of dyspareunia after menopause.*
4. Stable heterosexual partnership ≥2 years (or by investigator discretion if less than 2 years) and both partners want to have more satisfying penetrative intimacy.
5. No estrogen product use, local or systemic, for 6 months.*
6. More than 6 months of consistent insertional pain with intercourse (may have stopped having intercourse due to this consistent experience of pain).*
7. Willingness to enter a study where she will receive low-dose local estrogen.*
8. Willingness to enter a study that requires application of cream on a frequent schedule for 3 months. *
9. Willingness to evaluate the progress of therapies by use of the Tampon Test as many as 2 times per week, and willingness to attempt intercourse if the Tampon Test indicates tolerable penetrative pain.*

   * n/a for reference group

Exclusion Criteria:

1. Consistently has pain in the pelvis or low abdomen during or after intercourse (deep dyspareunia).
2. Negative cotton-swab touch test in the vulvar vestibule or vestibular tenderness that is not extinguishable by application of lidocaine 4% topical solution applied for 3 minutes.
3. Partner with sexual dysfunction limiting his performance or making it inconsistent. (The use of male therapy for erectile dysfunction is acceptable.)
4. Diagnosis by a physical therapist or clinician of significant pelvic floor muscle tension causing pain (pelvic floor myalgia) or has been found on screening examination to have pelvic floor tenderness or bladder tenderness.
5. Constant burning pain localized to the vulva.
6. Allergy to local estrogen products or lidocaine numbing agents.
7. Previous estrogen receptor positive breast cancer or endometrial cancer.
8. Endometrial thickness ≥5mm on screening via transvaginal ultrasound.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Goetsch, MD, MPH, Principal Investigator — Oregon Health & Science University, Portland, OR
Locations (1):
- Oregon Health & Science Univerity, Portland, Oregon, United States

REFERENCES:
- [Derived] Goetsch MF, Garg B, Lillemon J, Clark AL. Treating where it hurts-a randomized comparative trial of vestibule estradiol for postmenopausal dyspareunia. Menopause. 2023 May 1;30(5):467-475. doi: 10.1097/GME.0000000000002162. Epub 2023 Feb 14. PMID 36787525
- [Derived] Goetsch MF, Garg B, Lillemon J, Clark AL. Where does postmenopausal dyspareunia hurt? A cross-sectional report. Menopause. 2022 Jun 1;29(6):646-653. doi: 10.1097/GME.0000000000001956. PMID 35231008

RESULTS

PARTICIPANT FLOW:
Groups:
- 50mcg Estradiol Cream: Subjects randomized to 50mcg of study medication will be issued a pump that will dispense 0.5gm of cream with each pump
  50mcg estradiol cream: Use of study drug nightly
Period: Overall Study
Arm/Group | 50mcg Estradiol Cream | 100mcg Estradiol Cream
Started | 25 | 25
Completed | 25 | 22
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50mcg Estradiol Cream | 100mcg Estradiol Cream | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.24 (6.16) | 60.17 (7.7) | 59.69 (6.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 24 | 48
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: One was not analyzed because she was found to have a disqualifying diagnosis after the trial had commenced 1 mo.
  kg/m^2
    number analyzed (Participants) | 25 | 24 | 49
    (all) | 24.59 (4.04) | 25.91 (7.7) | 25.23 (4.61)

OUTCOME MEASURES:

1. Primary Outcome: Change in Median Dyspareunia Pain Scores After 4 Weeks Using Study Drug
Description: Change in median dyspareunia pain scores between baseline and 4 weeks of use of nightly use of study medication. Pain will be assessed using 11-point Numerical Rating Scale (NRS) where 0 = no pain and 10 = worst possible pain.
Time Frame: Baseline to 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50mcg Estradiol Cream | 100mcg Estradiol Cream
Number analyzed (Participants) | 25 | 22
score on a scale | -1.5 [-2 to -1] | -3 [-5 to -2]
Statistical Analysis 1: Comparison: 50mcg Estradiol Cream vs 100mcg Estradiol Cream; Test type: Non-Inferiority — We set 2 points (20%) as the margin of difference when defining and evaluating non-inferiority in comparing the 2 arms at 4 weeks; p = 0.08, Wilcoxon (Mann-Whitney) — Threshold for significance < 0.05; Median Difference (Final Values) = 2

2. Primary Outcome: Change in Median Pain Scores for Intercourse After 12 Weeks Using Study Drug
Description: Difference in median dyspareunia pain scores between arms for intercourse at 12 weeks after use of nightly study medication for 90d. Pain will be assessed using 11-point Numerical Rating Scale (NRS) where 0 = no pain and 10 = worst possible pain.
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50mcg Estradiol Cream | 100mcg Estradiol Cream
Number analyzed (Participants) | 25 | 22
score on a scale | -4 [-6 to -3] | -5.5 [-6 to -4.5]
Statistical Analysis 1: Comparison: 50mcg Estradiol Cream vs 100mcg Estradiol Cream; Test type: Non-Inferiority — We set 2 points (20%) as the margin of difference when evaluating non-inferiority in comparing the 2 arms at 4 weeks; p = 0.95, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2

ADVERSE EVENTS:
Time Frame: 3 months
Description: We assessed certain symptoms that could be potentially related to the intervention by including relevant questions on a questionnaire administered repeatedly through the intervention period.
Arm/Group | 50mcg Estradiol Cream | 100mcg Estradiol Cream
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 13/25 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mcg Estradiol Cream (N=25) | 100mcg Estradiol Cream (N=25)
mastalgia (Reproductive system and breast disorders) | 5 (7) | 3 (3)
increased headaches (Nervous system disorders) | 4 (4) | 4 (4)
increased hot flashes (Endocrine disorders) | 8 (9) | 5 (6)
postcoital spotting (Reproductive system and breast disorders) | 2 (2) | 0 (0)
local skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
fatigue (General disorders) | 0 (0) | 2 (2)
URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) — Cold
Candida vaginitis (Reproductive system and breast disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The design did not include a placebo arm. Therefore the various minor "adverse events" or side effects that were tabulated cannot be compared to the same complaints in a placebo arm. "Adverse events" includes specific possible estrogen side effects which were queried in repeating questionnaires rather than being volunteered by participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT03240081/Prot_SAP_000.pdf